CLINICAL TRIAL: NCT03926559
Title: The Effect of Neuraxial Morphine (Duramorph) on Pain Control
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1313375-3
Record Dates: First submitted 2019-01-08; First posted 2019-04-24 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Perineal Tear
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duramorph (Morphine) (Experimental): 2mg of Neuraxial Morphine given through epidural once after the patient has delivered.
  Interventions: Drug: Morphine.
- No intervention (No Intervention): Patient does not get any intervention.

INTERVENTIONS:
Drug: Morphine. — Pregnant patients with a perineal tear postpartum receive 2mg of morphine through their epidural. This will be a one time dose immediately postpartum.
  Other Names: Duramorph
  Arms: Duramorph (Morphine)

SUMMARY:
With the rise of the opioid epidemic, it is important for physicians to be more mindful of the amount of narcotic prescriptions that are being written every day. In the early postpartum period, pain and fatigue are the most common problems reported by women. Untreated pain has negative consequences on the amount of opioid narcotics used, postpartum depression, and the potential development of persistent chronic pain. While pain can interfere with a woman's ability to adequately take care of her newborn, narcotic abuse can lead to excessive maternal drowsiness and increased infant mortality in the new breastfeeding mother. The most common sources of pain after a vaginal delivery include breast engorgement, uterine contractions and perineal lacerations. Perineal lacerations are immediate postpartum complications of the vaginal birth process, defined as injury that involves the bulbocavernosum muscle complex (second degree), and may involve the anal sphincter complex (third degree) or the anal epithelium (fourth degree). Prevention of chronic and severe postpartum pain, especially after a cesarean delivery has been extensively studied, however, much paucity in research exists for the management of postpartum pain from perineal tears. Compared to patients with first degree tears or intact perineum, women with severe perineal lacerations (second degree or greater) have increased analgesic requirement up to the fifth postpartum day. . Epidural morphine has been accepted by anesthesiologists as treatment for acute pain. In obstetrics, 2-3 mg of epidural morphine was found to be sufficient to provide post-episiotomy analgesia. Neuraxial morphine has been used for analgesic management after a cesarean section, especially to reduce the amount of oral pain medications used in the first 24 hours, but limited data exists on the use of neuraxial morphine after a severe perineal laceration repair in the setting of a vaginal delivery. Niv et al (1994) studied the effect of epidural morphine and monitored its timing of administration in post-epiostomy pain onset. They noted that if epidural morphine is administered before the onset of pain in an episiotomy repair it is much more effective than if given after the onset. This study hopes to take the prior 1994 study a step further and incorporates it's data to investigate whether neuraxial morphine given after a severe perineal laceration repair mitigates postpartum pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a second degree, third degree, or fourth degree perineal tear identified in the immediate postpartum period.
* Pregnant patients who received neuraxial anesthesia during their labor course
* Women >18 yo

Exclusion Criteria:

* Unwillingness to participate in the study
* Allergy to morphine
* Women with history of polysubstance abuse/narcotic abuse
* Women <18 yo

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females
Enrollment: 125 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-21 (Estimated); Study Completion 2021-05-21 (Estimated)

PRIMARY OUTCOMES:
Postpartum pain | 24 hours postpartum
  Pain is to be assessed using the Numeric Rating Scale. Scale ranges from 1(no pain) to 10 (most pain). This scale will be used at 24 hours.
Delayed postpartum pain | 48 hours postpartum
  Pain is to be assessed using the Numeric Rating Scale. Scale ranges from 1(no pain) to 10 (most pain). This scale will be used at 48 hours to assess for delayed postpartum pain.

SECONDARY OUTCOMES:
Amount of narcotics used | 24 hours postpartum
  The number of narcotics will be calculated using the medical record number of the participant and by noting the narcotics that the patients received in a 24 hour time frame. This is documented by the nursing staff.
Amount of narcotics used | 48 hours postpartum
  The number of narcotics will be calculated using the medical record number of the participant and by noting the narcotics that the patients received in a 48 hour time frame. This is documented by the nursing staff.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University Medical Center, North Augusta, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No